CLINICAL TRIAL: NCT04260971
Title: Cyclic Versus Continuous Deep Brain Stimulation in Essential Tremor
Brief Title: Cyclic Deep Brain Stimulation in Essential Tremor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KCH20-025; 270731 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Deep Brain Stimulation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 2 groups with either cyclical or continuous stimulation. Patients will cross-over to the 2nd mode of stimulation after 1 month and then continued on the preferred mode of stimulation for the 3rd month. Open label follow-up starts at this point and continues for another 9 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study adopts a blind design. Only the programmer is aware of the randomisation details and the parameters will be kept separately in order to keep others blind about the intervention. Unblinding of the study will occur at the 3rd month of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclical Stimulation (Experimental): This group will undergo cyclical stimulation mode of stimulation
  Interventions: Device: Abbott St Jude Medical Infinity 7 neurostimulator
- Continuous Stimulation (Active Comparator): This group will undergo the standard continuous mode of stimulation
  Interventions: Device: Abbott St Jude Medical Infinity 7 neurostimulator

INTERVENTIONS:
Device: Abbott St Jude Medical Infinity 7 neurostimulator — The stimulator has the capability to deliver both continuous and cyclical modes of stimulation which is being investigated in this study

SUMMARY:
The aim of the study is to prove the efficacy and safety of cyclical deep brain stimulation (DBS) in patients with essential tremor, and demonstrate non-inferiority of cyclical DBS on tremor control when compared to continuous stimulation.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind cross-over trials. Patients will be randomized into two groups in a cross-over fashion to have either continuous or cyclical stimulation for a total of three months. Following this, the trial will be unblinded and open-label follow up will continue for another nine months. Device use as per standard practice continues after the end of the trial.

If the hypothesis is proven correct, this will provide proof of concept that cyclical stimulation for the treatment of essential tremor results in improved battery life, reduced number of operations for battery changes, reduction in stimulation side-effects and enhancing quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is at least 18 years of age
2. Participant has confirmed diagnosis of medically-refractory essential tremor
3. Participant meets criteria for implantation of DBS system
4. Participant understands the study requirements and treatments procedures and provides informed consent before any study-specific tests or procedures are performed

Exclusion Criteria:

1. Participant meets any contraindications for implantation of DBS system
2. Participant is undergoing or has had previous thalamic stimulation either in a research trial or with a permanent implant
3. Participant is unwilling or unable to comply with all study required follow-up evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Fahn-Tolosa-Marin Tremor Rating Scale - total score difference | 6 months compared to baseline
  Change in Fahn-Tolosa-Marin tremor rating scale at 6 months compared to baseline. Minimum score is 0 and maximum score is 84. Higher scores indicate worse tremor control

SECONDARY OUTCOMES:
EuroQol five dimensions questionnaire (EQ-5D) difference | 6 months post activation compared to baseline
  The total score of EQ-5D questionnaire at 6 months compared to baseline. Each dimension of the questionnaire has a minimum score of 1 and a maximum score of 5. Higher composite scores indicate increased levels of perceived problems
Beck's Depression Index questionnaire difference | 6 months post activation compared to baseline
  The total score of Beck's Depression Index questionnaire at 6 months compared to baseline. The minimum score is 0 and maximum score is 63. Higher scores indicate increasing severity of depression
Quality of Life in Essential Tremor (QUEST) questionnaire difference | 6 months post activation compared to baseline
  The total score of Quality of Life in Essential Tremor questionnaire at 6 months compared to baseline. Minimum score is 0 and maximum score is 120 with higher scores indicating worse quality of life due to tremor
Satisfaction with Treatment (SWT) questionnaire difference | 6 months post activation compared to baseline
  The difference in Satisfaction with Treatment outcomes at 6 months compared to baseline
Clinical Global Impression of Change (CGI) difference | 6 months post activation compared to baseline
  The difference in Clinical Global Impression of change outcome at 6 months compared to baseline
Implantable Pulse Generator (IPG) power consumption and longevity | 6 months compared to baseline
  Total amount of implantable pulse generator consumption used compared between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Keyoumars Ashkan, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira JJ, Mestre TA, Lyons KE, Benito-Leon J, Tan EK, Abbruzzese G, Hallett M, Haubenberger D, Elble R, Deuschl G; MDS Task Force on Tremor and the MDS Evidence Based Medicine Committee. MDS evidence-based review of treatments for essential tremor. Mov Disord. 2019 Jul;34(7):950-958. doi: 10.1002/mds.27700. Epub 2019 May 2. PMID 31046186
- [Background] Flora ED, Perera CL, Cameron AL, Maddern GJ. Deep brain stimulation for essential tremor: a systematic review. Mov Disord. 2010 Aug 15;25(11):1550-9. doi: 10.1002/mds.23195. PMID 20623768
- [Background] Koller WC, Lyons KE, Wilkinson SB, Troster AI, Pahwa R. Long-term safety and efficacy of unilateral deep brain stimulation of the thalamus in essential tremor. Mov Disord. 2001 May;16(3):464-8. doi: 10.1002/mds.1089. PMID 11391740
- [Background] Rehncrona S, Johnels B, Widner H, Tornqvist AL, Hariz M, Sydow O. Long-term efficacy of thalamic deep brain stimulation for tremor: double-blind assessments. Mov Disord. 2003 Feb;18(2):163-70. doi: 10.1002/mds.10309. PMID 12539209
- [Background] Wharen RE Jr, Okun MS, Guthrie BL, Uitti RJ, Larson P, Foote K, Walker H, Marshall FJ, Schwalb J, Ford B, Jankovic J, Simpson R, Dashtipour K, Phibbs F, Neimat JS, Stewart RM, Peichel D, Pahwa R, Ostrem JL; SJM DBS ET Study Group. Thalamic DBS with a constant-current device in essential tremor: A controlled clinical trial. Parkinsonism Relat Disord. 2017 Jul;40:18-26. doi: 10.1016/j.parkreldis.2017.03.017. Epub 2017 Mar 30. PMID 28400200
- [Background] Paschen S, Forstenpointner J, Becktepe J, Heinzel S, Hellriegel H, Witt K, Helmers AK, Deuschl G. Long-term efficacy of deep brain stimulation for essential tremor: An observer-blinded study. Neurology. 2019 Mar 19;92(12):e1378-e1386. doi: 10.1212/WNL.0000000000007134. Epub 2019 Feb 20. PMID 30787161
- [Background] Hariz GM, Blomstedt P, Koskinen LO. Long-term effect of deep brain stimulation for essential tremor on activities of daily living and health-related quality of life. Acta Neurol Scand. 2008 Dec;118(6):387-94. doi: 10.1111/j.1600-0404.2008.01065.x. Epub 2008 Jul 8. PMID 18616684
- [Background] Troster AI, Pahwa R, Fields JA, Tanner CM, Lyons KE. Quality of life in Essential Tremor Questionnaire (QUEST): development and initial validation. Parkinsonism Relat Disord. 2005 Sep;11(6):367-73. doi: 10.1016/j.parkreldis.2005.05.009. PMID 16103000